CLINICAL TRIAL: NCT04810208
Title: A Phase Ia/Ib, First-in-human, Open Label, Multicentre, Dose-escalation and Dose-expansion Study of a Novel NanoZolid®-Docetaxel Depot Formulation (NZ-DTX Depot) Given as an Intra-tumoural Injection in Patients With Advanced Solid Tumours
Brief Title: Intratumoural Injection of a Novel NanoZolid®-Docetaxel Depot Formulation in Patients With Advanced Solid Tumours
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic decision
Sponsor: Lidds AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NZ-DTX-001
Record Dates: First submitted 2021-03-18; First posted 2021-03-22 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NZ-DTX Depot (Experimental)
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Docetaxel — Docetaxel in NanoZolid formulation, for intratumoural injection

SUMMARY:
This is a multicentre, open-label, first in man, study of a novel NanoZolid®-docetaxel depot formulation (NZ-DTX Depot) given as an intra-tumoural injection in patients with advanced solid tumours. The study includes a dose escalation part and a dose expansion part.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent granted before undertaking any study-specific procedures;
2. Male or female patient ≥18 years of age on the day of consenting to the study;
3. Histologically or cytologically confirmed diagnosis of solid cancer;
4. At least 1 advanced solid, palpable, cutaneous or subcutaneous tumour lesion with following characteristics:

   * a cutaneous lesion with of thickness ≥4 mm and diameter ≥25 mm at the longest axis, or
   * a subcutaneous lesion of diameter ≥20 mm at the longest and the shortest axis;
5. Eastern Co-operative Oncology Group (ECOG) performance status (PS) 0-2;
6. Patient from one the following categories:

   * Patient for whom no standard therapy exists, or standard therapy is contraindicated, or
   * Patient who is scheduled for other anti-cancer treatment (e.g. radiotherapy, immunological treatment, surgery) which will start after completion of at least one treatment cycle of NZ-DTX, i.e after the end-of-study (EOS) visit.

Exclusion Criteria:

1. Known hypersensitivity to any of the excipients in the NZ-DTX Depot formulation (docetaxel, calcium sulphate, sodium carboxymethylcellulose);
2. Life expectancy <3 months;
3. Bleeding deficiencies or ongoing anticoagulant therapy that would put the patient at increased risk of clinically significant bleeding, in the judgement of the Investigator. If the patient has an international normalised ratio (INR) below 1.2 the Investigator may judge if interruption of anticoagulant therapy is warranted;
4. Any of the following abnormal laboratory values at screening;

   * Bone marrow function:

     * Absolute neutrophil count (ANC) <1.5 x 109/l;
     * Platelet count <100 x 109/l;
     * Haemoglobin <9.0 mg/dl.
   * Coagulation:

     - International Normalized Ratio (INR) >1.2.
   * Hepatic, renal, and biochemistry parameters:

     * Aspartate transaminase (AST) or alanine transaminase (ALT) >2.5 x upper limit of normal (ULN) (>5 x ULN if liver metastases present)*;
     * Alkaline phosphatase (ALP) >2.5 x ULN;
     * Total bilirubin >1.5 x ULN;
     * Estimated glomerular filtration rate (eGFR) <40 ml/min/1.73 m² using the Modified Cockcroft & Gault formula.

       * For patients with liver impairment who have serum transaminase levels (ALT and/or AST) greater than 1.5 times x ULN - the doses will be restricted to max. 75mg/m2. In the event this is not possible the patient will not be included.
5. Severe fluid retention, e.g. pulmonary oedema, pleural effusion, pericardial effusion or ascites;
6. Clinically significant heart disease (i.e. heart failure or myocardial infarction within 6 months of screening, instable angina pectoris);
7. History of thromboembolic or cerebrovascular events within 6 months of screening;
8. Major surgery within 2 weeks of screening, or patient not recovered from major surgery;
9. Known untreated or uncontrolled acute infection, including urinary tract infection, within 7 days of screening;
10. Not recovered from Grade 2 or higher adverse events (AEs) due to previous treatments, excepting alopecia;
11. Concurrent participation in another investigational study;
12. Last investigational drug administration in a prior investigational study within 14 days of study treatment initiation or <5 times the half-life of the investigational drug, whichever is longer;
13. Last administration of other anti-neoplastic drug within 14 days of study treatment initiation;
14. Radiotherapy of lesion to be injected within 4 weeks of first treatment with NZ-DTX Depot, or irradiated lesion to be injected without signs of disease progression since irradiation;
15. For men and women of childbearing potential: Unwillingness to follow contraception requirements;
16. Female patients with planned or current pregnancy and/or currently breastfeeding;
17. Any other severe, acute or chronical medical or psychiatric condition or laboratory abnormality that, in the judgement of the Investigator, would make the patient inappropriate for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2021-10-07 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of NZ-DTX Depot given as an intra-tumoural injection in solid, palpable, cutaneous or subcutaneous tumour lesions. | 5 weeks
  The MTD will be determined by incidence of DLTs
The recommended Phase 2 dose (RP2D) of NZ-DTX Depot given as an intra-tumoural injection in a solid, palpable cutaneous or subcutaneous tumour lesion. | 5 weeks
  The RP2D will be determined by frequency and severity of adverse events

SECONDARY OUTCOMES:
Frequency and severity of treatment-emergent adverse events [safety and tolerability] following an intratumoural injection of NZ-DTX Depot | 5 weeks
  Frequency and severity of treatment-emergent adverse events
Plasma concentration of docetaxel, following an intratumoural injection of NZ-DTX Depot | 5 weeks
  Plasma concentration of docetaxel
Anti-tumour effect following an intratumoural injection of NZ-DTX Depot | 5 weeks
  Tumour response by RECIST

OTHER OUTCOMES:
Presence of immune biomarkers in plasma, following an intratumoural injection of NZ-DTX Depot | 9 weeks
  Analysis of cytokines in plasma
Presence of immune biomarkers in tissue, following an intratumoural injection of NZ-DTX Depot | 9 weeks
  Immunohistochemistry analysis [PD-L1] in tissue

CONTACTS AND LOCATIONS:
Overall Officials: Charlotta Gauffin, PhD, Study Director — Lidds AB
Locations (4):
- Herlev Hospital, Copenhagen, Denmark
- Lithuania (2):
  - Lithuanian University of Health Sciences, Kaunas
  - National Cancer Institute, Vilnius
- Karolinska University Hospital, Stockholm, Sweden